CLINICAL TRIAL: NCT04532762
Title: Demonstration of a Decongestant Effect of "Coldamaris Akut" Compared to Saline Nasal Spray in Subjects Suffering From Grass Pollen Induced Rhinitis/Rhinoconjunctivitis.
Brief Title: Demonstration of a Decongestant Effect of "Coldamaris Akut" Compared to Saline Nasal Spray.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COA_19_03
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-08

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
Keywords: Allergic Rhinoconjunctivitis; Allergic Rhinitis; Coldamaris akut; Vienna Challenge Chamber; Nasal Congestion Symptom; Carrageenan; Carragelose; Iota-carrageenan
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: This is a prospective, placebo-controlled, double-blinded randomized two-way cross-over single site study in adult subjects (18 to 65 years) who demonstrate a grass pollen specific Immunoglobulin E (IgE) reactivity and have a history of grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma. In the cross-over setting Coldamaris akut nasal spray will be evaluated compared to Coldamaris sine 0.5% nasal spray.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coldamaris akut (Experimental): One puff (140µl) into each nostril
  Interventions: Device: nasal spray
- Placebo (Placebo Comparator): One puff (140µl) into each nostril
  Interventions: Device: nasal spray

INTERVENTIONS:
Device: nasal spray — Application of a nasal spray

SUMMARY:
Allergic rhinitis (AR) in its seasonal and perennial form is a common allergic condition. The majority of allergic rhinitis sufferers report nasal (congestion, sneezing, itching and rhinorrhea) and ocular (redness, watery eyes, itching and burning) symptoms.

Coldamaris akut nasal spray is a Carragelose® containing hyperosmolar solution that is indicated for supportive treatment in case of blocked nose due to rhinitis of any kind. Carragelose® is a sulfated polymer from red seaweed also widely used in the food industry and has GRAS status (FDA). The increased osmolality is based on the addition of sorbitol. This clinical study has the aim to show that Coldamaris akut has a mild decongestant effect.

This will be a prospective, controlled, double-blinded randomized two-way cross-over single site study in adult subjects (18 to 65 years) who demonstrate a grass pollen specific Immunoglobulin E (IgE) reactivity and have a history of grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma. In the cross-over setting two treatments, namely Coldamaris Akut and Coldamaris sine will be evaluated.

The objective of the trial is to demonstrate a decongestant effect on the nasal mucosa of patients treated with Coldamaris akut nasal spray compared to subjects treated with Coldamaris sine nasal spray in grass pollen induced rhinitis/rhinoconjunctivitis.

The evaluation will be based on the assessment of nasal congestion symptom during grass pollen challenge performed in the Vienna Challenge Chamber (environmental exposure chamber).

Secondary objective of the trial is to demonstrate the clinical performance of Coldamaris akut nasal spray on nasal symptoms compared to subjects treated with saline nasal spray.

DETAILED DESCRIPTION:
This is a prospective, placebo-controlled, double-blinded randomized two-way cross-over single site study in adult subjects (18 to 65 years) who demonstrate a grass pollen specific Immunoglobulin E (IgE) reactivity and have a history of grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma. In the cross-over setting Coldamaris akut nasal spray will be evaluated compared to Coldamaris sine nasal spray.

Visit 1 - Screening:

At least one week prior to first treatment block, subjects will be screened for appropriate allergic response. A total nasal symptom score (TNSS) of at least 6 points out of 12 with a single symptom score for "nasal congestion" ≥ 2 within the first two hours in the grass pollen challenge chamber is required to be included into the study. If a screening for appropriate allergic response was done during the last 6 months, results from this allergy challenge can be used to fulfil the respective inclusion criteria.

Visit 2 - Inclusion:

In addition to the screening provocation the medical and allergic history, safety lab as well as retrieving inclusion and exclusion criteria will be assessed via anamnesis. Furthermore, all safety assessments will be conducted.

Note: Visit 1 and visit 2 could be done on the same day!

Visit 3: Day1 of first treatment period Eligible subjects will be randomly assigned to one of the two treatment arms (fully blinded) in the order of appearance and their screening numbers assigned at visit 1. Subjects will enter the study site about one hour ahead of the start of allergen provocation. After positive completion of all study relevant assessments, subjects will be randomized and enter the allergy challenge chamber for 6 hours. About one hour forty-five minutes after entry (after the eighth subjective score), the first treatment with the respective nasal spray will take place under staff supervision.

The subjective nasal symptom score will be recorded every fifteen minutes during a 6-hour allergen exposure challenge. Anterior rhinomanometry will be performed regularily.

Visit 4: Day1 of second treatment period Subjects will enter the study site about one hour ahead of the start of allergen provocation. In the following Visit 4 will be done in the same way as Visit 3.

Between the respective study treatments, a wash-out period of at least 7 days must be adhered to allowing complete symptom relief from previous challenge. After the wash-out period, subjects change to the second treatment block.

During the entire trial, subjects will be asked to monitor for adverse events (AEs), and they will record the use of concomitant medications on the provided form.

One week after the final provocation session, subjects will complete the trial after their follow up visit.

The trial design is appropriate for the indication studied. Validated methods of data collection, analysis, and evaluation will be used for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed
* Healthy male or female subjects aged 18 to 65 years
* A documented clinically relevant allergic history of moderate to severe SAR to grass pollen for the previous two years
* Subjects exhibit a moderate to severe response to approximately 1500 grass pollen grains/m3 within the first 2 hours in the Vienna Challenge Chamber, which is defined as total nasal symptom score (TNSS) of at least 6 (out of 12) with the necessity to score at least "moderate = 2" for the single symptom "nasal congestion" using standard VCC grass pollen allergen mixture. Nasal symptom score is the sum of "nasal congestion", "rhinorrhea", "itchy nose" and "sneezing", each of which have been scored on a categorical scale from 0 to 3.
* Positive Skin Prick Test (SPT) response (wheal diameter at least 3 mm larger than diluent control) to grass pollen SPT solutions (standard Allergopharma) at screening or within the last 12 months prior to study start.
* Positive serum specific IgE against recombinant major allergen components of the used grass pollen e.g. g6 (specific CAP IgE ≥0.70 kU/L) at screening or within the last 12 months prior to study start.
* Asthma patients only if the asthma condition is mild or intermittent, and if those are not treated with steroids
* Subject has a forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value (ECCS) at the screening.
* Subject is capable of understanding the study procedures and potential risks associated with the study, and voluntarily agrees to participate by giving written informed consent.
* Subject is able to adhere to dose and visit schedules.
* Subject is able to read, understand and complete questionnaires and diaries.

Exclusion Criteria:

* A clinical history of uncontrolled asthma within 3 months prior to screening
* Subjects with asthma requiring treatment with inhaled corticosteroids on a regular basis judged by the
* investigator
* Previous successful immunotherapy to grass pollen, a grass pollen allergen or a cross-reacting allergen within the past 3 years
* Ongoing treatment with any allergen-specific immunotherapy product
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other
* relevant infectious process at randomisation
* Clinically relevant nasal polyps, medical history of paranasal sinus surgery and/or medical history of surgery of
* nasal turbinates judged by the investigator
* Subjects using any ophthalmic steroids during the last 30 days
* Subjects treated with nasal, inhaled or systemic steroids during the last 30 days
* History of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise induced, food allergy, drugs
* or an idiopathic reaction)
* Any clinically relevant chronic disease judged by the investigator
* Systemic disease affecting the immune system judged by the investigator
* Use of an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to screening
* History of allergy, hypersensitivity or intolerance to any ingredients of the study medication
* History of alcohol or drug abuse.
* Being immediate family of the investigator or trial staff, defined as the investigator's/staff's spouse, parent, child,grandparent or grandchild
* Subjects treated with leukotriene antagonists (1 month before study start), long-lasting anti-histamines, like
* cetirizine, fexofenadine, loratadine, desloratadine, hydroxyzine (5 to 10 days before study start), mast cell
* stabilizer (2 weeks before study start) or nasal decongestant (3 days before study start)
* Subjects with an acute or chronic sinusitis judged by the investigator
* Positive Serology result judged by the investigator
* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted and safe birth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Nasal Congestion Symptom Score (NCSS) | 0-6 hourse of allergen exposure challenge
  calculated as the baseline adjusted mean of NCSS measured every 15 minutes during the grass pollen allergen exposure challenge from time-point 0 to 6 hours.
  The NCSS is scored on a 4-point scale from 0-3 with "0"= none "1"=mild "2"=moderate "3"=severe

SECONDARY OUTCOMES:
Nasal airflow | 0-6 hourse of allergen exposure challenge
  will be assessed every 30 minutes during the six hour grass pollen allergen exposure challenge; an additional assessment takes place at timepoint 2:15
Total nasal symptom score (TNSS) | 0-6 hourse of allergen exposure challenge
  Total nasal symptom score (TNSS) is the sum of the symptoms "nasal congestion", "rhinorrhea", "itchy nose","sneezing".
  Each individual symptom of TNSS will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe).
Total ocular symptom score (TOSS) | 0-3 hourse of allergen exposure challenge
  Total ocular symptom score (TOSS) is the sum of the symptoms "ocular itching", "redness", "watery eyes".
  Each individual symptom of TOSS will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe). TOSS will be assessed every 15 minutes during the three hour grass pollen allergen exposure challenge.
Total asthma symptom score (TASS) | 0-3 hourse of allergen exposure challenge
  Total asthma symptom score (TASS) is the sum of the symptoms "cough", "wheeze", "dyspnea".
  Each individual symptom of TASS will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe). TASS will be assessed every 15 minutes during the three hour grass pollen allergen exposure challenge.
Nasal secretion | 0-6 hourse of allergen exposure challenge
  will be assessed every 30 minutes during the six hour grass pollen allergen exposure challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prieschl-Grassauer, PhD, Study Chair — CSO
Locations (1):
- Vienna Challenge Chamber, Vienna, Austria

REFERENCES:
- [Derived] Unger-Manhart N, Morokutti-Kurz M, Zieglmayer P, Russo A, Siegl C, Konig-Schuster M, Koller C, Graf P, Graf C, Lemell P, Savli M, Zieglmayer R, Dellago H, Prieschl-Grassauer E. Decongestant Effect of "Coldamaris Akut", a Carrageenan- and Sorbitol-Containing Nasal Spray in Seasonal Allergic Rhinitis. Int J Gen Med. 2024 Nov 8;17:5105-5121. doi: 10.2147/IJGM.S476707. eCollection 2024. PMID 39534593